CLINICAL TRIAL: NCT03210311
Title: Determining the Role of Pre-existing Factors, Early Diagnostic Options and Early Treatment in the Development of Breast Cancer Related Lymphedema
Brief Title: Pre-existing Factors, Early Detection and Early Treatment of Breast Cancer Related Lymphedema
Acronym: DEARLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, dr. Sarah Thomis, Vascular Surgeon, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S60382; 2017-002306-12 (EudraCT Number)
Record Dates: First submitted 2017-06-29; First posted 2017-07-06 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Lymphedema of Upper Arm; Breast Cancer; Diagnoses Disease
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): * Receive information: the patient receive a leaflet with information about the lymphatic system and lymphedema, clinical evaluation and conservative treatment of lymphedema
  * Perform skin care
  * Perform twice a day upper limb exercises at home. They are advised to use the arm as normal as possible.
- intervention group (Active Comparator): * Receive information: the patient receive a leaflet with information about the lymphatic system and lymphedema, clinical evaluation and conservative treatment of lymphedema
  * Perform skin care
  * Perform upper limb exercises at home twice a day. They are advised to use the arm as normal as possible
  * Wear a compression sleeve
  Interventions: Device: compression

INTERVENTIONS:
Device: compression — a compression stocking is worn, a garment compression class 2, flat knitted
  Arms: intervention group

SUMMARY:
Breast-cancer related lymphoedema (BCRL) is a common phenomenon. Early diagnosis and treatment is very important to alter the normal progression of this disease. A threshold (>= 3% volume change) that recognizes subclinical lymphedema is promoted. When the lymphedema is diagnosed late, options for treatment are diminished as fibrous tissue is formed.

Preoperative investigation with near-infrared fluorescence lymphography can show an abnormality. Even if a linear transport is visualized, velocity of the transport can be diminished or a different pathway than normal can be visualized. Such an extensive evaluation has not been performed yet.

This lymphofluoroscopy gives an opportunity to detect lymphedema earlier than clinically visible (subclinical). The investigators hypothesize that the evolution of lymphedema can be altered if treatment is started in the subclinical phase.

DETAILED DESCRIPTION:
Breast-cancer related lymphoedema (BCRL) is a common phenomenon. Estimates of incidence rates have varied over time, especially since the progression to less invasive techniques as sentinel node procedures and radiotherapy. According to a review article of DiSipio the incidence of arm lymphedema was about four times higher in women who had an axillary lymph node dissection (18 studies; 19.9%, 13.5-28.2) than in those who had sentinel lymph node biopsy (18 studies; 5.6%, 6.1-7.9). Several other risk factors are already suggested as having a negative impact on the development of lymphedema such as BMI and chemotherapy. A comprehensive overview of all treatment related risk factors and patient related risk factors, including demographics, has not been reported yet.

Lymphedema is identified with upper limb volume measurements eg circumference measurements, water displacement and perometer. Bioimpedance spectroscopy can also be used to assess the extracellular fluid. A 10% limb volume change has been reported as the most accurate threshold to diagnose lymphedema. However, with this definition an underestimation of the incidence rate of lymphoedema is made. Therefore, recently a threshold of 5% limb volume change is proposed.

A study by Rockson et al suggested that in almost 75 % of the cases, lymphoedema is established in the first year after breast cancer treatment. But up to two years after surgery, there still is a possibility to develop lymphoedema.

Early diagnosis and treatment is very important to alter the normal progression of this disease. A threshold (>= 3% volume change) that recognizes subclinical lymphedema is promoted.

When the lymphedema is diagnosed late, options for treatment are diminished as fibrous tissue is formed.

During near-infrared fluorescence lymphography (lymphofluoroscopy), a fluorescent substance is injected subcutaneously in the hand and the transport of lymph is visualized from the hand up to the axilla. A normal transport is defined as a linear image and an abnormal transport as a dermal backflow image. The dermal backflow image is divided in three different classifications according to the severity.

Preoperative investigation with near-infrared fluorescence lymphography can show an abnormality. Even if a linear transport is visualized, velocity of the transport can be diminished or a different pathway than normal can be visualized. Such an extensive evaluation has not been performed yet.

This lymphofluoroscopy gives an opportunity to detect lymphedema earlier than clinically visible (subclinical).

The investigators hypothesize that the evolution of lymphedema can be altered if treatment is started in the subclinical phase.

ELIGIBILITY:
Inclusion Criteria:

* Age >18y (since the investigation using ICG is not dangerous for pregnant women, women with child bearing age are included)
* Women/ men with breast cancer and scheduled for unilateral axillary lymph node dissection (ALND) or sentinel node biopsy (SNB)
* Oral and written approval of informed consent
* Dutch speaking

Exclusion Criteria:

* Oedema of the upper limb from other causes
* Cannot participate during the entire study period
* Mentally or physically unable to participate in the study
* Contra-indication for the use of ICG: allergy to iodine, hyperthyroidism
* Metastatic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Incidence of lymphedema of arm and hand | up to 36 months
  defined as 5% volume increase compared to the contralateral side
Deterioration of dermal backflow | up to 36 months
  measured by lymphofluoroscopy

SECONDARY OUTCOMES:
Change of extracellular fluid change of extracellular fluid | up to 36 months
  measured by the BIS
Change of quality of life | up to 36 months
  measured by Mc Gill questionnaire
change of pitting status | up to 36 months
  measured by the pitting test at each visit
Change of water content | up to 36 months
  measured with moisture meter
change of skinfold tickness | up to 36 months
  measured by skinfold
relative change of arm volume difference | up to 36 months
  relative volume difference at assessment - relative volume difference at baseline
severity of disturbance of lymphatic transport | up to 36 months
  scoring dermal backflow in the 13 regions
problems in functioning related to development of lymphedema | up to 36 months
  measured by lymph ICF questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Thomis, MD, Principal Investigator — UZ Leuven
Locations (1):
- Vascular surgey Lymphovenous center, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomis S, Devoogdt N, Bechter-Hugl B, Nevelsteen I, Neven P, Fourneau I. Impact of a compression garment, on top of the usual care, in patients with breast cancer with early disturbance of the lymphatic transport: protocol of a randomised controlled trial. BMJ Open. 2020 Dec 4;10(12):e042018. doi: 10.1136/bmjopen-2020-042018. PMID 33277289